CLINICAL TRIAL: NCT02885740
Title: Role and Interactions of Adenosine, Receptors, Methionine Cycle Nutritional, Metabolic and Genetic Determinants in the Onset of Atrial Fibrillation in Normal Heart
Acronym: FACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-A01197-50
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atrial fibrillation in normal heart (Experimental): Patients having atrial fibrillation in normal heart
  Interventions: Other: Quantification assay of adenosine and methionine cycle metabolites; Genetic: Polymorphism analysis of genes related to adenosine metabolism and methionine cycle; Other: Quantitative and qualitative nutritional evaluation; Biological: Blood sample
- Control (Active Comparator): Patients having a junctional supraventricular tachycardia in normal heart
  Interventions: Other: Quantification assay of adenosine and methionine cycle metabolites; Genetic: Polymorphism analysis of genes related to adenosine metabolism and methionine cycle; Other: Quantitative and qualitative nutritional evaluation; Biological: Blood sample

INTERVENTIONS:
Other: Quantification assay of adenosine and methionine cycle metabolites
Genetic: Polymorphism analysis of genes related to adenosine metabolism and methionine cycle
Other: Quantitative and qualitative nutritional evaluation — Questionnaire on consumption of 208 foods and drinks
Biological: Blood sample

SUMMARY:
The purpose of this study is to analyze the association of atrial fibrillation onset in normal heart and:

* Genetic determinants (genes of receptors, enzymes involved in synthesis and degradation, genes of bioavailability of coenzymes and nutritional precursors)
* Metabolic determinants of adenosine and methionine cycles
* Nutritional determinants.

Secondary purposes are:

* Analysis of physiopathologic mechanisms of AF in normal hearts and adenosine metabolisms and its interaction with methionine metabolism, according to identified genetic determinants
* Analysis of blood markers of adenosine and methionine metabolites as phenotypic markers of detected polymorphisms
* Evaluate the role of adenosine receptors in AF onset

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most frequent arrhythmia and its causes are not well known. Experimental and clinical studies showed that activation of parasympathetic system can induce and maintain AF. Adenosine is a cardiovascular modulator with effects on vascular tonus and activation of nodal tissue through the activation of A1, A2A, A2B et A3 receptors. Intracellular production of adenosine is directly dependent (30%) on the hydrolysis of S-adenosylhomocysteine (SAH) by S-adenosylhomocysteine hydrolase in methionine cycle. Cellular production of adenosine depends on ratio SAH/S-adenosylmethionine (SAM) and modulates the expression of receptors. Other potential interactions between this 2 metabolisms in AF are: 1) ratio SAM/SAH influences epigenetic mechanisms that can modify the expression of candidate genes involved in synaptic transmission and potassium canals, 2) ratio SAM/SAH influences also the cellular production of homocysteine with effects on cellular polarization, 3) adenosine and homocysteine are factors involved in thrombophilia and potentially associated to thromboembolic complications of AF.

This study will evaluate the genetic (micro SNP-array) and adenosine and methionine metabolic determinants in the physiopathology of AF in normal hearts.

Perspectives of this study are the prevention of AF in normal hearts through a nutritional and metabolic approach in subjects having a multigenic predisposition.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Affiliation to French social security plan

AF in normal heart:

- Atrial fibrillation in normal heart

Control:

- Junctional supraventricular tachycardia in normal heart

Normal heart: absence of macroscopic cardiomyopathy (echocardiography and normal ejection fraction)

Exclusion Criteria:

* Considerable consumption of coffee (> 50 mg/day, 15 cups/day)
* Actual administration of drugs interfering with adenosine metabolism: dipyridamole and methotrexate
* Actual administration interfering with methionine metabolism: folates, methotrexate and anticonvulsants
* Known renal insufficiency
* Known hypo- or hyperthyroidism
* Refusal or impossibility of informed consent
* Pregnant or breastfeeding women
* Person deprived of liberty
* Person under legal protection or not able to consent
* Person in emergency situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-03; Primary Completion 2017-01 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of genetic polymorphisms related to adenosine and methionine metabolism | day 0
  Increase of frequency in patients having an AF in normal heart
Levels of adenosine and methionine cycle nutritional and metabolic determinants | day 0

SECONDARY OUTCOMES:
Level of nutritional and methionine cycle metabolic determinants according to thromboembolic complications of AF in normal heart | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Etienne ALIOT, Pr, Principal Investigator — Département de Cardiologie, CHU Nancy, Hôpitaux de Brabois, France
Locations (1):
- Département de Cardiologie, CHU Nancy, Hôpitaux de Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No